CLINICAL TRIAL: NCT02045264
Title: An Open-label, Single-arm Study to Assess the Pharmacokinetics, Safety, and Tolerability of a Single Subcutaneous Dose of Icatibant in Healthy Japanese Volunteers
Brief Title: Open-label, Single-arm Study to Assess the Pharmacokinetics, Safety, and Tolerability of a Single Subcutaneous Dose of Icatibant in Healthy Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP-FIR-101
Record Dates: First submitted 2014-01-13; First posted 2014-01-24 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Firazyr; Angioedema; Angioedemas, Hereditary; Vascular Diseases; Cardiovascular Diseases; Urticaria; Skin Diseases, Vascular; Skin Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Genetic Diseases, Inborn; Icatibant; Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Non-Narcotic; Analgesics; Sensory System Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Pharmacologic Actions; Anti-Inflammatory Agents; Therapeutic Uses; Antirheumatic Agents; Adrenergic beta-Antagonists; Adrenergic Antagonists; Adrenergic Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; Central Nervous System Agents
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema; Vascular Diseases; Cardiovascular Diseases; Urticaria; Skin Diseases, Vascular; Skin Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Genetic Diseases, Inborn | interventions — icatibant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Icatibant (30 mg) (Experimental): 30mg dose of icatibant is administered as a single subcutaneous injection in the abdominal area
  Interventions: Drug: Icatibant (30 mg)

INTERVENTIONS:
Drug: Icatibant (30 mg) — On Day 1, subjects will receive a single 30mg subcutaneous injection of icatibant in their abdominal area. Subjects will be discharged from the study on Day 3 after collection of study related assessments
  Other Names: Firazyr

SUMMARY:
This is a single-dose study to evaluate the pharmacokinetics, safety, and tolerability of icatibant administered to adult Japanese subjects.

DETAILED DESCRIPTION:
Icatibant has been studied for the treatment of acute attacks of hereditary angioedema (HAE), an autosomal dominant disorder characterized by recurrent and self-limiting episodes of edema of the skin, larynx, and gastrointestinal tract. The most serious manifestation of an HAE attack is laryngeal edema, causing obstruction of the upper airways that may lead to death by asphyxiation if undiagnosed and/or untreated.

Icatibant has been approved in over 40 countries around the world including the United States (US) and Europe for the treatment of acute attacks of hereditary angioedema (HAE) in adults. This study is being conducted to evaluate the safety and tolerability of icatibant in a Japanese population and to evaluate whether race/ethnicity impacts the pharmacokinetics of icatibant after single subcutaneous injection.

This is an open-label, single-arm study that will enroll at least 12 Japanese subjects (in order to have 12 subjects complete the study), age 18-55 years inclusive. All subjects will receive a single subcutaneous injection of 30mg icatibant. The study will be conducted at 1 site in the US. The study will consist of a Screening Period, a Treatment Period, and a Follow-Up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers, 18 to 55 years of age, inclusive; healthy status defined as absence of clinically significant findings in medical history or screening assessments
2. Japanese; defined as born in Japan, lived outside of Japan for no more than 10 years, and having Japanese parents and Japanese maternal and paternal grandparents
3. Body mass index of 18 to 28 kg/m2, inclusive

Exclusion Criteria:

1. History of, or current, clinically significant disease and/or abnormalities
2. Smoking habit in excess of 5 cigarettes per day or the equivalent within 30 days of Day 1 or inability to refrain from smoking during the study confinement period
3. Subject has current abnormal thyroid function, as defined as abnormal screening thyroid stimulating hormone (TSH) and free thyroxine (T4). Treatment with a stable dose of thyroid medication for at least 12 weeks is permitted
4. History of drug allergy or other allergy that, in the opinion of the investigator, contraindicates participation
5. Male subjects who consume more than 21 units of alcohol per week or 3 units per day. Female subjects who consume more than 14 units of alcohol per week or 2 units per day. (1 alcohol unit =1 beer or =1 wine (5oz/150mL) or =1 liquor (1.5oz/40mL) or =0.75oz alcohol)
6. Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches. (1 caffeine unit is contained in the following items: one 6oz (180mL) cup of coffee, two 12oz (360mL) cans of cola, one 12oz cup of tea, three 1oz (85g) chocolate bars. Decaffeinated coffee, tea, or cola are not considered to contain caffeine)
7. Current use of any medication (including over-the-counter, herbal, or homeopathic preparations) with the exception of female hormonal replacement therapy or hormonal contraceptives. Occasional use of over-the-counter doses of ibuprofen or acetaminophen for minor self-limited pain (eg, headaches) is also acceptable. Current use is defined as use within 7 days of the first dose of investigational product\
8. Pregnant or lactating females

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2014-02-27 (Actual); Study Completion 2014-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- PAREXEL, Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Icatibant (30 mg): Subjects received a 30mg dose of icatibant administered as a single subcutaneous injection in the abdominal area on Day 1.
Period: Overall Study
Arm/Group | Icatibant (30 mg)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set consisted of all subjects who had taken the single dose of icatibant.
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of Icatibant and Metabolites
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: Over 48 hours post-dose
Population: The Pharmacokinetic Set consisted of all subjects who had taken the single dose of icatibant and for whom the primary pharmacokinetic data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
ng/mL
  Icatibant | 1190 (261)
  Metabolite 1 | 340 (67.7)
  Metabolite 2 | 365 (74.8)

2. Primary Outcome: Time to Peak Plasma Concentration (Tmax) of Icatibant and Metabolites
Description: Tmax is the time after administration of a drug when the maximum plasma concentration in the body is reached.
Time Frame: Over 48 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
hr
  Icatibant | 0.67 (0.20)
  Metabolite 1 | 1.92 (0.289)
  Metabolite 2 | 1.92 (0.289)

3. Primary Outcome: Drug Concentration Half-Life (T1/2) of Icatibant and Metabolites
Description: The time it takes for the blood plasma concentration of a substance to halve.
Time Frame: Over 48 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
hr
  Icatibant | 1.77 (0.356)
  Metabolite 1 | 3.69 (0.579)
  Metabolite 2 | 4.11 (1.01)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUCinf) of Icatibant and Metabolites
Description: AUCinf is the area under the plasma concentration versus time curve extrapolated from time 0 to infinity, calculated using the observed value of the last non-zero concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Over 48 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
ng*hr/mL
  Icatibant | 2320 (403)
  Metabolite 1 | 1750 (308)
  Metabolite 2 | 1960 (346)

5. Primary Outcome: Total Body Clearance (CL/F) of Icatibant
Description: The rate at which a drug is removed from the body.
Time Frame: Over 48 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
mL/hr | 13200 (1890)

6. Secondary Outcome: The Total Number of Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) were those that started after the single dose of icatibant.
Time Frame: TEAEs were collected after the single dose of icatibant until follow up, 5-7 days after icatibant administration
Population: The Safety Set consisted of all subjects who had taken the single dose of icatibant.
Measure: Number; unit: Treatment Emergent Adverse Events
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
Treatment Emergent Adverse Events | 2

7. Secondary Outcome: The Percentage of Subjects With Any Injection Site Reactions.
Time Frame: Over 48 hours post-dose
Population: The Safety Set consisted of all subjects who had taken the single dose of icatibant.
Measure: Number; unit: percentage of participants
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
percentage of participants
  Erythema | 100.00
  Warm sensation | 50.00
  Swelling | 91.67
  Cutaneous pain | 33.33
  Itching/Pruritus | 8.33
  Burning sensation | 8.33

8. Secondary Outcome: Safety Evaluation Measured by Percentage of Subjects With Not Clinically Significant Abnormalities in ECG Results
Time Frame: Over 48 hours post-dose
Population: The Safety Set consisted of all subjects who had taken the single dose of icatibant.
Measure: Number; unit: percentage of participants
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
percentage of participants
  Screening | 91.67
  Day 1, Pre-dose | 50.00
  Baseline | 50.00
  Day 1, 0.75 hours | 33.33
  Day 1, 8 hours | 33.33
  Day 2, 24 hours | 66.67
  Day 3, 48 hours | 66.67

9. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Icatibant and Metabolites
Description: AUC0-t is the area under the plasma concentration versus time curve extrapolated from time 0 to to the last quantifiable concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Over 48 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
ng*hr/mL
  Icatibant | 2320 (402)
  Metabolite 1 | 1740 (307)
  Metabolite 2 | 1950 (345)

10. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Time Frame: Over 48 hours post-dose
Population: The Safety Set consisted of all subjects who had taken the single dose of icatibant.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
mmHg
  Day 1, 0.5 h | -2.0 (6.42)
  Day 1, 1 h | -3.8 (4.30)
  Day 1, 2 h | -5.2 (4.57)
  Day 1, 4 h | -5.2 (7.52)
  Day 1, 6 h | -4.8 (8.07)
  Day 1, 8 h | -4.5 (6.67)
  Day 1, 12 h | -3.4 (9.06)
  Day 2, 24 h | -1.8 (7.76)
  Day 3, 48 h | -5.3 (6.18)

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Time Frame: Over 48 hours post-dose
Population: The Safety Set consisted of all subjects who had taken the single dose of icatibant.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
mmHg
  Day 1, 0.5 h | -1.8 (12.07)
  Day 1, 1 h | -1.9 (13.03)
  Day 1, 2 h | -5.8 (14.21)
  Day 1, 4 h | -7.3 (17.06)
  Day 1, 6 h | -4.3 (16.20)
  Day 1, 8 h | -3.0 (11.52)
  Day 1, 12 h | -4.4 (14.11)
  Day 2, 24 h | -6.2 (11.98)
  Day 3, 48 h | -6.4 (12.72)

12. Secondary Outcome: Change From Baseline in Pulse Rate
Time Frame: Over 48 hours post-dose
Population: The Safety Set consisted of all subjects who had taken the single dose of icatibant.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Icatibant (30 mg)
Number analyzed (Participants) | 12
beats per minute
  Day 1, 0.5 h | 1.4 (7.53)
  Day 1, 1 h | 0.1 (5.38)
  Day 1, 2 h | -3.0 (9.67)
  Day 1, 4 h | -6.3 (9.91)
  Day 1, 6 h | -0.1 (11.15)
  Day 1, 8 h | -3.6 (10.88)
  Day 1, 12 h | -3.2 (10.50)
  Day 2, 24 h | -6.8 (9.02)
  Day 3, 48 h | -4.0 (9.77)

ADVERSE EVENTS:
Arm/Group | Icatibant (30 mg)
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icatibant (30 mg) (N=12)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Injection Site Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.